CLINICAL TRIAL: NCT06668311
Title: The Impact of Play Dough and Picture Books on Physiological Parameters, Anxiety, and Fear in 3-6-Year-Old Children During Nebulizer Treatment: a Randomized Controlled Study
Brief Title: Play Dough and Picture Books: Reducing Anxiety and Fear in 3-6-Year-Olds During Nebulizer Treatment
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Responsible Party: Principal Investigator, Ilcim Ercan Koyuncu, Lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Nebulizer Treatment
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Nebulizer Therapy
Keywords: nursing care; nubulizer therapy; pediatric emergency department

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Play Dough Group (Experimental): The child will be provided with play dough five minutes before the commencement of nebulizer treatment and will be allowed to continue playing with it throughout the treatment.
  Interventions: Other: play dough
- Picture Book Reading group (Experimental): Five minutes before the commencement of nebulizer treatment, the child will be provided with a picture book and will be allowed to continue reading it throughout the treatment.
  Interventions: Other: picture book reading
- Control Group (No Intervention): Nebulizer treatment of the child will be performed by the routine protocols currently applied in the emergency department.

INTERVENTIONS:
Other: play dough — 1. Children and families will be informed about the purpose of the study and their verbal and written consent will be obtained.
  2. The first part of the Patient Information Form will be completed for children who accept the study.
  3. The second part of the Patient Information Form will be completed five minutes before nebulizer treatment.
  4. Five minutes before nebulizer treatment, play dough will be given to the child.
  5. The child will be allowed to play with the play dough during the nebulizer treatment.
  6. The second part of the Patient Information Form will be filled in at the 5th minute of the treatment and after the treatment is over.
  7. The application will take approximately 15 minutes.
  Arms: Play Dough Group
Other: picture book reading — 1. Children and families will be informed about the purpose of the study and their verbal and written consent will be obtained.
  2. The first part of the Patient Information Form will be completed for children who accept the study.
  3. The second part of the Patient Information Form will be completed five minutes before nebulizer treatment.
  4. Five minutes before nebulizer treatment, the child will be given a picture book.
  5. Picture book will be read to the child during the treatment.
  6. The second part of the Patient Information Form will be filled in at the 5th minute of the treatment and after the treatment is over.
  7. The application will take approximately 15 minutes.
  Arms: Picture Book Reading group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of play dough and picture books on physiological parameters, anxiety, and fear levels in children aged 3-6 undergoing nebulizer treatment. The trial will involve two groups: an intervention group engaging with play dough and picture books during treatment and a control group receiving standard care. Physiological data, including heart rate and oxygen saturation, will be monitored alongside behavioral assessments of anxiety and fear. This study seeks to determine whether these non-pharmacological interventions can alleviate distress in young children, contributing to more child-friendly treatment approaches in pediatric healthcare.

ELIGIBILITY:
Inclusion Criteria:

* Being in the 3-6 age group
* Follow-up in the emergency department with upper or lower respiratory tract disease
* Application of nebuliser therapy
* Staying with the parent during the research
* To be able to speak and understand Turkish
* Parents' consent to participate in the study

Exclusion Criteria:

* Having a disease that causes maladaptive behaviours (ADHD, Autism, etc.)
* Having a chronic disease affecting the respiratory tract
* Chronic diseases or serious infections affecting vital signs
* Implementation of droplet or contact isolation
* Having a physical disability that will prevent him/her from playing with playdough
* Having a cognitive disability that prevents reading books

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-11-15 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Fear | 5 minutes before the treatment, at the beginning of treatment, 5th minutes into the treatment, immediately after the treatment
  The scale was developed for the age group of 4-10 years and is used in studies up to 3 years of age. It consists of five facial expressions ranging from neutral (0 points: no anxiety) to frightened face (4 points: severe anxiety). The child is asked to mark the degree of fear by choosing the most appropriate facial expression. As the score obtained from the scale increases, the child's level of fear increases.
Anxiety | 5 minutes before the treatment, at the beginning of treatment, 5th minutes into the treatment, immediately after the treatment
  The scale is in the form of a thermometer. The bottom part of the thermometer is labelled as 'Calm: Not tense or anxious (0 points)', and the top part is rated as "Very tense or anxious (10 points)". To assess the child's state of anxiety, the child is asked to mark how he/she feels 'right now' on the thermometer. As the score obtained from the scale increases, the anxiety level of the child increases.

SECONDARY OUTCOMES:
Pulse Rate | 5 minutes before the treatment, at the beginning of treatment, 5th minutes into the treatment, immediately after the treatment
  Maintaining and normalizing pulse rate within normal range (75-115 per minute)
Respiratory Rate | 5 minutes before the treatment, at the beginning of treatment, 5th minutes into the treatment, immediately after the treatment
  Maintaining and normalizing respiratory rate within normal range (20-25 per minute)
Saturation rate | 5 minutes before the treatment, at the beginning of treatment, 5th minutes into the treatment, immediately after the treatment
  Maintaining and normalizing saturation rate within normal range (95-100%)

CONTACTS AND LOCATIONS:
Locations (1):
- Başkent University, Ankara, Beşevler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goralski JL, Davis SD. Breathing easier: addressing the challenges of aerosolizing medications to infants and preschoolers. Respir Med. 2014 Aug;108(8):1069-74. doi: 10.1016/j.rmed.2014.06.004. Epub 2014 Jun 25. PMID 25012949
- [Background] Esposito-Festen J, Ijsselstijn H, Hop W, van Vliet F, de Jongste J, Tiddens H. Aerosol therapy by pressured metered-dose inhaler-spacer in sleeping young children: to do or not to do? Chest. 2006 Aug;130(2):487-92. doi: 10.1378/chest.130.2.487. PMID 16899849
- [Background] Erzinger S, Schueepp KG, Brooks-Wildhaber J, Devadason SG, Wildhaber JH. Facemasks and aerosol delivery in vivo. J Aerosol Med. 2007;20 Suppl 1:S78-83; discussion S83-4. doi: 10.1089/jam.2007.0572. PMID 17411409
- [Background] DiBlasi RM. Clinical Controversies in Aerosol Therapy for Infants and Children. Respir Care. 2015 Jun;60(6):894-914; discussion 914-6. doi: 10.4187/respcare.04137. PMID 26070582
- [Background] Supat B, Brennan JJ, Vilke GM, Ishimine P, Hsia RY, Castillo EM. Characterizing pediatric high frequency users of California emergency departments. Am J Emerg Med. 2019 Sep;37(9):1699-1704. doi: 10.1016/j.ajem.2018.12.015. Epub 2018 Dec 12. PMID 30651182
- [Background] Durak H, Uysal G. The Effect of Cartoon Watching and Distraction Card on Physiologic Parameters and Fear Levels During Inhalation Therapy in Children: A Randomized Controlled Study. J Trop Pediatr. 2021 Jan 29;67(1):fmab018. doi: 10.1093/tropej/fmab018. PMID 33742204
- See also: Related Info — https://iris.who.int/bitstream/handle/10665/356584/9789240051140eng.pdf?sequence=1
- See also: Related Info — https://data.tuik.gov.tr/Bulten/Index?p=Turkiye-Saglik-Arastirmasi-2022-49747
- See also: Related Info — https://www.aarc.org/wp-content/uploads/2018/01/aerosol-guide-for-hcp-3rd.pdf